CLINICAL TRIAL: NCT05684458
Title: The Effect of Reiki on Symptom Control and Quality of Life in Breast Cancer Patients: A Randomized Controlled Trial
Brief Title: The Effect of Reiki on Symptom Control and Quality of Life in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, NURSEMIN UNAL, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 114
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Symptoms and Signs; Quality of Life
Keywords: Reiki; breast cancer; symptom control; quality of life
MeSH Terms: conditions — Breast Neoplasms; Signs and Symptoms | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The patients and the investigators know which group they are assigned to. Only the outcome assessor doesn't know which patient is assigned to which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki Group (Experimental): Patient Descriptive Information Form, Edmonton Symptom Diagnosis Scale (ESTO), and European Association for Cancer Research and Treatment BR23 Quality of Life Scale (EORTC-QLQ-BR232) will be administered to the Reiki group. Then, under the guidance of a researcher holding a Usui Reiki Master & Teacher degree, a total of 26 patients in the intervention group will be given a short 30-minute application to energy centers by researchers with a second-degree Reiki practitioner. On the second and on third days, 30 minutes of short Reiki will be done remotely. After 3 days and 10 days after the patients were included in the study, the post-tests will be performed by calling the patients.
  Interventions: Procedure: Reiki
- Control Group (No Intervention): Patient Descriptive Information Form, Edmonton Symptom Diagnosis Scale (ESTO), and European Association for Cancer Research and Treatment BR23 Quality of Life Scale (EORTC-QLQ-BR232) will be administered to the control group. No treatment will be applied to the patients. Post-tests will be applied to all patients 3 days and 10 days after they were included in the study.

INTERVENTIONS:
Procedure: Reiki — Reiki, a non-invasive, free and safe complementary therapy method, is practiced with a series of hand positions held on the patient's body to help balance the life force energy.
  Arms: Reiki Group

SUMMARY:
The aim of this study is to examine the effect of Reiki on symptom control and quality of life in breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the world's second most common type of cancer, the most frequently diagnosed cancer in women, and the leading cause of cancer death. Energy therapies have an essential place in complementary and alternative treatments that are commonly used in breast cancer patients. Reiki, practiced by trained practitioners, is performed by activating the body's energy centers, including blood and lymph circulation, and stimulating the nervous system, thus providing energy circulation and providing mental-physical relaxation, positively affecting health. The effect of Reiki on cancer patients has been shown in studies that it can relieve pain, reduce anxiety and depression, improve quality of life and reduce fatigue.

In this study, women with stage 3 and 4 metastatic breast cancer who were diagnosed with breast cancer for at least 3 months and received at least two cycles of chemotherapy in the outpatient chemotherapy unit of the Medical Oncology outpatient clinic of a training and research hospital will be included. It is aimed to reach a total of 52 women who meet the inclusion criteria and agreed to participate in the study between February 1, 2023, and July 30, 2023. Patient Descriptive Information Form, Edmonton Symptom Diagnosis Scale (ESTO), and European Association for Cancer Research and Treatment BR23 Quality of Life Scale (EORTC-QLQ-BR232) preliminary tests will be applied to all women. Patients will be randomized 1:1 into groups by a single therapist according to the block randomization method. Under the guidance of a researcher holding a Usui Reiki Master & Teacher degree, a total of 26 patients in the intervention group will be given a short 30-minute application to energy centers by researchers with a second-degree Reiki practitioner. On the second and on third days, 30 minutes of short Reiki will be done remotely. No treatment will be applied to 26 patients in the control group. Post-tests will be applied to all patients 3 days and 10 days after they were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women with at least 3 months of breast cancer diagnosis, at least two cycles of chemotherapy, and stage 3 and 4 metastatic breast cancer.

Exclusion Criteria:

* Those who have difficulty in responding to the data collection form to be used in the research and have problems in understanding and communicating Turkish,
* Those who refuse to answer the Reiki application and data collection tools,
* Those who want to leave the research while the research is continuing,
* Those who received any supplementary application in the last 6 months will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients with breast cancer will be included in the study.
Enrollment: 52 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient Descriptive Information Form | Baseline
  The form created by the researchers included 11 questions covering the sociodemographic and medical characteristics.
Change from Edmonton Symptom Diagnosis Scale | Change from baseline Edmonton Symptom Diagnosis Scale at 3rd days and 10th days
  It was developed by Bruera et al. in 1991. Ten symptoms are questioned as pain, fatigue, nausea, sadness, anxiety, insomnia, loss of appetite, well-being, shortness of breath and other problems. In the Turkish validity and reliability study of the scale, 3 additional symptoms (changes in the skin and nails, sores in the mouth, numbness in the hands) were added to the other problems section in line with the literature information. The patient is asked to match his symptoms with a number that he thinks is most suitable for him from the numbers from 0 to 10. The number 0 indicates no symptoms, the number 10 indicates that the symptom is very severe. Pre-chemotherapy Cronbach α value of ESAS was 0.83; Cronbach's α ESAS after chemotherapy is 0.76.
Change from European Association for Cancer Research and Treatment BR23 Quality of Life Scale | Change from baseline European Association for Cancer Research and Treatment BR23 Quality of Life Scale at 3rd days and 10th days
  The scale is a quality of life scale specially prepared for breast cancer by the European Cancer Research and Treatment Organization. It can be applied to all breast cancer patients, regardless of the stage of the disease and the treatment method. Its Turkish validity and reliability were evaluated by Demirci et al. in 2011. and the Cronbach alpha value was found to be 0.90. This scale is divided into two subgroups as functional and symptom scales. Scoring is made as 1 (none)-4 (very much). Higher functional dimension scores indicate higher quality of life. A high score in the symptoms dimension indicates a low quality of life, and low scores indicate a high quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nursemin Unal, Principal Investigator — Ankara Medipol University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steinhorn DM, Din J, Johnson A. Healing, spirituality and integrative medicine. Ann Palliat Med. 2017 Jul;6(3):237-247. doi: 10.21037/apm.2017.05.01. Epub 2017 May 22. PMID 28595441
- [Background] Bruera E, Kuehn N, Miller MJ, Selmser P, Macmillan K. The Edmonton Symptom Assessment System (ESAS): a simple method for the assessment of palliative care patients. J Palliat Care. 1991 Summer;7(2):6-9. PMID 1714502
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Ong'udi M, Mutai P, Weru I. Study of the use of complementary and alternative medicine by cancer patients at Kenyatta National Hospital, Nairobi, Kenya. J Oncol Pharm Pract. 2019 Jun;25(4):918-928. doi: 10.1177/1078155218805543. Epub 2018 Oct 14. PMID 30319064
- [Background] Frisch N, Butcher HK, Campbell D, Weir-Hughes D. Holistic Nurses' Use of Energy-Based Caring Modalities. J Holist Nurs. 2018 Sep;36(3):210-217. doi: 10.1177/0898010116665447. Epub 2016 Sep 1. PMID 27587296
- [Background] Buyukbayram Z, Citlik Saritas S. The effect of Reiki and guided imagery intervention on pain and fatigue in oncology patients: A non-randomized controlled study. Explore (NY). 2021 Jan-Feb;17(1):22-26. doi: 10.1016/j.explore.2020.07.009. Epub 2020 Jul 31. PMID 32778391